CLINICAL TRIAL: NCT02345863
Title: A Prospective, Open-label, Multicenter Phase-II Trial to Evaluate the Efficacy and Safety of a Sequential Regimen of Bendamustine Followed by GA101 and Ibrutinib (BIG) Followed by GA101 and Ibrutinib Maintenance in CLL Patients (CLL2-BIG Protocol)
Brief Title: Sequential Regimen of Bendamustin [B] Followed by GA101 and Ibrutinib [I] in CLL Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Collaborators: Hoffmann-La Roche (Industry); Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL2-BIG; 2014-000569-35 (EudraCT Number)
Record Dates: First submitted 2015-01-12; First posted 2015-01-26 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Chronic Lymphocytic Leucemia
Keywords: CLL
MeSH Terms: interventions — Bendamustine Hydrochloride; obinutuzumab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendamustine + GA101 + Ibrutinib (Experimental): Bendamustine 70mg/m² i´v
  GA101: 1000 mg iv
  Ibrutinib: 420 mg po daily
  Interventions: Drug: Bendamustine; Drug: GA101; Drug: Ibrutinib

INTERVENTIONS:
Drug: Bendamustine — Debulking:
  2 cycles of Bendamustine (70 mg/m² iv) will be administered before induction unless a contraindication is existing or it is not clinically indicated.
Drug: GA101 — Induction
  GA101 iv infusion:
  Cycle 1: Day 1 100 mg Day 1 (or 2) 900 mg Day 8 1000 mg Day 15 1000 mg Cycle 2-6: Day 1 1000 mg
  Maintenance After the induction ibrutinib po 420 mg daily and GA101 iv 1000 mg every three months will be continued.
  GA101: Cycle 1-8 Day 1 1000 mg
  Other Names: Obinutuzumab
Drug: Ibrutinib — Ibrutinib will be administered as a daily oral dosage of 420 mg starting on cycle 2 day 1.
  Cycle 2-6: Day 1 420 mg daily
  Maintenance After the induction ibrutinib po 420 mg daily and GA101 iv 1000 mg every three months will be continued.
  Ibrutinib: Cycle 1-8 420 mg daily

SUMMARY:
A prospective, open-label, multicenter Phase-II trial to evaluate the efficacy and safety of a sequential regimen of Bendamustine followed by GA101 and Ibrutinib followed by Ibrutinib and GA101 maintenance in CLL patients.

DETAILED DESCRIPTION:
In the CLL2-BIG trial an allcomer CLL population with indication for treatment will be included.

Patient will receive 2 cycles of debulking treatment with bendamustin unless contraindications are existing or debulking is not indicated.

Afterwards 6 cycles of induction therapy with GA101 and ibrutinib will be applied, each with a duration of 28 days. Primary endpoint overall Response rate will be assessed at final restaging.

Patients benefitting from BIG treatment will enter the maintenance phase of the trial. Maintenance treatment will be continued if no unacceptable toxicity occurs until three months after negativity of minimal residual disease [MRD] is achieved in peripheral blood in patients with (clinical) complete response (CR) or (clinical) incomplete complete response [CRi] (confirmed by 2 consecutive testings of MRD within 3 months), progression of CLL, start of a subsequent therapy or up to 8 cycles of maintenance (each cycle with a duration of 84 calendar days = 3 months), whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. documented CLL requiring treatment (irrespective if first- or relapse treatment) according to the criteria of the international Workshop of CLL [iwCLL]

   In case of previously treated patients, these must have recovered from acute toxicities and treatment regimen must be stopped within the following time periods before start of the study treatment in the CLL2-BIG trial:
   * chemotherapy within ≥ 28 days
   * antibody treatment within ≥ 14 days
   * kinase inhibitors, B-cell-lymphoma 2 [BCL2] -antagonists or immunomodulatory agents within ≥ 3 days
   * corticosteroids may be applied until the start of the BIG-regimen, these have to be reduced to an equivalent of ≤ 20mg prednisolon during treatment
2. Creatinine clearance ≥ 30 ml/min
3. Adequate hematologic function
4. Adequate liver function
5. Negative serological testing for hepatitis B, hepatitis-C RNA and negative HIV test within 6 weeks prior to registration
6. Age at least 18 years
7. Eastern Cooperative Oncology Group [ECOG] status 0 - 2; ECOG 3 is only permitted if related to CLL
8. Life expectancy ≥ 6 months
9. Ability and willingness to provide written informed consent and to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Transformation of CLL
2. Known central nervous system (CNS) involvement
3. Patients with a history of confirmed progressive multifocal leukoencephalopathy [PML]
4. Malignancies other than CLL currently requiring systemic therapies
5. Uncontrolled infection requiring systemic treatment
6. Use of investigational agents which would interfere with the study drug within 28 days prior to registration
7. Any comorbidity or organ system impairment rated with a cumulative illness rating scale [CIRS] score of 4, excluding the eyes/ears/nose/throat/larynx organ system or any other life-threatening illness, medical condition or organ system dysfunction that - in the investigator´s opinion could comprise the patients safety or interfere with the absorption or metabolism of the study drugs (e.g, inability to swallow tablets or impaired resorption in the gastrointestinal tract)
8. Known hypersensitivity to GA101, ibrutinib or any of the excipients
9. Requirement of treatment with strong cytochrome P450 3A4 [CYP3A4] -inhibitors/-inducers or anticoagulant with warfarin or phenprocoumon (marcumar)
10. History of stroke or intracranial hemorrhage within 6 months prior to registration
11. Pregnant women and nursing mothers
12. Fertile men or women of childbearing potential unless:surgically sterile or ≥ 2 years after the onset of menopause or willing to use two methods of reliable contraception including one highly effective (Pearl Index <1) and one additional effective (barrier) method during study treatment and for 18 months after end of study treatment.
13. Vaccination with a live vaccine a minimum of 28 days prior to registration
14. Legal incapacity
15. Prisoners or subjects who are institutionalized by regulatory or court order
16. Persons who are in dependence to the sponsor or an investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-01-16 (Actual); Primary Completion 2016-08-22 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 84 days after first dose of last induction cycle
  proportion of patients responding according to international working Group on chronic lymphocytic leukemia criteria

SECONDARY OUTCOMES:
Safety: Adverse events (AEs) and adverse events of special interest (AESI) | up to 48 months after first dose of study drug
  Type, frequency, and severity of adverse events (AEs) and adverse events of special interest (AESI) and their relationship to study treatment.
minimal residual disease (MRD) | final restaging and during maintenance
  Rate of MRD responses in peripheral blood measured by immunophenotyping

CONTACTS AND LOCATIONS:
Overall Officials: Julia von Tresckow, Dr. med., Principal Investigator — German CLL Study Group
Locations (1):
- German CLL Study Group, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] von Tresckow J, Cramer P, Bahlo J, Robrecht S, Langerbeins P, Fink AM, Al-Sawaf O, Illmer T, Klaproth H, Estenfelder S, Ritgen M, Fischer K, Wendtner CM, Kreuzer KA, Stilgenbauer S, Bottcher S, Eichhorst BF, Hallek M. CLL2-BIG: sequential treatment with bendamustine, ibrutinib and obinutuzumab (GA101) in chronic lymphocytic leukemia. Leukemia. 2019 May;33(5):1161-1172. doi: 10.1038/s41375-018-0313-8. Epub 2018 Dec 19. PMID 30568174
- [Derived] Langerbeins P, Giza A, Robrecht S, Cramer P, von Tresckow J, Al-Sawaf O, Fink AM, Furstenau M, Kutsch N, Simon F, Goede V, Hoechstetter M, Niemann CU, da Cunha-Bang C, Kater A, Dubois J, Gregor M, Staber PB, Tausch E, Schneider C, Stilgenbauer S, Eichhorst B, Fischer K, Hallek M. Reassessing the chronic lymphocytic leukemia International Prognostic Index in the era of targeted therapies. Blood. 2024 Jun 20;143(25):2588-2598. doi: 10.1182/blood.2023022564. PMID 38620092
- [Derived] Cramer P, Tausch E, von Tresckow J, Giza A, Robrecht S, Schneider C, Furstenau M, Langerbeins P, Al-Sawaf O, Pelzer BW, Fink AM, Fischer K, Wendtner CM, Eichhorst B, Kneba M, Stilgenbauer S, Hallek M. Durable remissions following combined targeted therapy in patients with CLL harboring TP53 deletions and/or mutations. Blood. 2021 Nov 11;138(19):1805-1816. doi: 10.1182/blood.2020010484. PMID 34086865